CLINICAL TRIAL: NCT05445908
Title: A Phase 2 Clinical Study of SKB264 With/Without KL-A167 in Patients With Unresectable Locally Advanced, Recurrent or Metastatic HER2-negative Breast Cancer Who Have Not Received Prior Systemic Therapy
Brief Title: SKB264 +/- KL-A167 in Recurrent or Metastatic HER2-negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅱ-07
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Triple-negative Breast Cancer and HR+/HER2- BC
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 18-O-demethylcervinomycin A2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SKB264+KL-A167（Part1，TNBC） (Experimental): Participants received SKB264 followed by KL-A167
  Interventions: Drug: SKB264; Drug: KL-A167
- SKB264（Part2，TNBC） (Experimental): Participants received SKB264
  Interventions: Drug: SKB264
- SKB264+KL-A167（Part2，TNBC） (Experimental): Participants received SKB264 followed by KL-A167
  Interventions: Drug: SKB264; Drug: KL-A167
- SKB264（Part3，HR+/HER2- BC） (Experimental): Participants received SKB264
  Interventions: Drug: SKB264
- SKB264+KL-A167（Part3，HR+/HER2- BC） (Experimental): Participants received SKB264 followed by KL-A167
  Interventions: Drug: SKB264; Drug: KL-A167

INTERVENTIONS:
Drug: SKB264 — SKB264 will be administered as an intravenous (IV) infusion every 2 weeks on Day 1 of each 14-day cycle
Drug: KL-A167 — KL-A167 will be administered as an intravenous (IV) infusion every 2 weeks on Day 1 of each 14-day cycle
  Arms: SKB264+KL-A167（Part1，TNBC）; SKB264+KL-A167（Part2，TNBC）; SKB264+KL-A167（Part3，HR+/HER2- BC）

SUMMARY:
The purpose of this study is to assess the safety and tolerability and preliminary antitumor activity of SKB264 with/without KL-A167 in patients with unresectable locally advanced, recurrent or metastatic TNBC and HR+/HER2- BC .The study is divided into three parts.Part 1（TNBC）: exploratory phase of the efficacy and safety of the combination treatment. Part 2（TNBC）: The subjects will be randomized to treatment group for SKB264 + KL-A167 or SKB264 . Part 3（HR+/HER2- BC）: The subjects will be randomized to treatment group for SKB264 + KL-A167 or SKB264 .

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 and ≤ 75 years at the time of signing the informed consent form (ICF);
2. Histological and/or cytological diagnosis of TNBC or HR+/HER2- BC based on pathology reports on recent biopsy samples or other pathological samples (central laboratory confirmation is not required)；
3. Patients have not received prior systemic chemotherapy for locally advanced, recurrent and metastatic disease；
4. Ability to provide fresh or archival tumor tissue for biomarker testing and analysis;
5. Patients with at least one measurable lesion per RECIST v1.1 criteria, and patients with only skin or bone lesions cannot be enrolled;
6. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 with an expected survival of ≥ 12 weeks;
7. Adequate organ and bone marrow function;
8. Patients must recover from all toxicities due to prior treatment (recovery to ≤ Grade 1 based on CTCAE v5.0 assessment, or meeting the inclusion criteria in the protocol) with the exception of alopecia and vitiligo;
9. Female subjects of childbearing potential and male patients with partners of childbearing potential who use effective medical contraception during the study treatment period and for 6 months after the end of dosing (see Appendix for specific contraceptive measures);
10. Patients voluntarily participate in the study, sign the ICF, and will be able to comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

1. History of other malignancies;
2. Patients with a history of central nervous system (CNS) metastases or current CNS metastases.
3. Imaging (CT or MRI) shows that the tumor has invaded large blood vessels or the investigator judges that the tumor is likely to invade important blood vessels and cause fatal hemorrhage during the follow-up study；
4. Received any systemic immune-stimulatory agents within 4 weeks prior to the first dose of study; Received any traditional Chinese medicine for approved anti-tumor indications within 2 weeks prior to the first dose of study;
5. Received other clinical investigational drugs within 4 weeks or major surgery within 4 weeks prior to the first dose of the study treatment;
6. Patients who required systemic corticosteroids (> 10 mg/day prednisone or equivalent; low-dose corticosteroids are allowed, such as ≤10 mg/day prednisone or equivalent, if the dose is stable for 4 weeks), or other immunosuppressive therapy within 2 weeks prior to the first dose. Steroids are allowed as prophylaxis for hypersensitivity reactions;
7. Patients who occurred arteriovenous thrombosis within 6 months prior to the first dose of study treatment，Such as cerebrovascular accidents, deep vein thrombosis, and pulmonary embolism, etc.
8. Prior treatment with a TROP2-targeted drug or checkpoint inhibitor ;
9. Serious or uncontrolled cardiac disease or clinical symptoms requiring treatment；
10. Patients with (noninfectious) interstitial lung disease (ILD) or history of pneumonia requiring steroid therapy; patients with serious pulmonary function impairment due to lung disease;
11. Uncontrolled systemic disease as judged by the investigator, included uncontrolled hypertension, uncontrolled diabetes, pesence of pleural effusion, pericardial effusion, or ascites that is clinically symptomatic or requires repeated drainage;
12. Active autoimmune disease requiring systemic treatment within the past 2 years;
13. Active hepatitis B or hepatitis C; known history of positive human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS); positive syphilis antibody test;
14. Known hypersensitivity to the study drug or any of its components, or severe allergic reactions to other monoclonal antibodies;
15. Pregnant or lactating women;
16. Any patient whose condition deteriorates rapidly during the screening process prior to the first dose, such as severe changes in performance status, unstable pain requiring adjustment of analgesic therapy, etc;
17. Other circumstances that, in the opinion of the investigator, are not appropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From baseline up to 30 days after last dose or to the beginning of the new anti-cancer therapy, up to 24 months
  Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Objective Response Rate (ORR) | From baseline to first documented objective response, up to 24 months
  Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR), assessed by Investigator based on RECIST version 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From baseline to the first documented disease progression or date of death (whichever occurs first), up to 24 months
  Progression-free survival (PFS) was defined as the time from baseline to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause. PD was defined as at least a 20% increase in the sum of diameters of target lesions.
Duration of response (DOR) | From the date of first objective response (CR or PR) to the date of first documentation of PD or death (whichever occurs first), up to 24 months
  Duration of Response (DOR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. DoR was measured for responding subjects (PR or CR) only.
Disease control rate (DCR) | From baseline to date of first documented objective response (CR, PR, and SD), up to 24 months
  Disease control rate (DCR) was defined as the sum of complete response (CR) rate, partial response (PR) rate, and stable disease (SD) rate. As per RECIST v1.1, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) of SKB264-ADC, SKB264-TAB and free KL610023 | Cycles 1-3, 5, 7, 9, and 11, every 6 cycles starting from Cycle 17 Day 1: pre-dose, post-dose (each cycle is 14 days), up to 24 months
Pharmacokinetic Parameter Minimum Plasma Concentration (Cmin) of SKB264-ADC, SKB264-TAB and free KL610023 | Cycles 1-3, 5, 7, 9, and 11, every 6 cycles starting from Cycle 17 Day 1: pre-dose, post-dose (each cycle is 14 days), up to 24 months
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) of KL-A167 | Cycles 1-3, 5, 7, 9, and 11, every 6 cycles starting from Cycle 17 Day 1: pre-dose, post-dose (each cycle is 14 days), up to 24 months
Pharmacokinetic Parameter Minimum Plasma Concentration (Cmin) of KL-A167 | Cycles 1-3, 5, 7, 9, and 11, every 6 cycles starting from Cycle 17 Day 1: pre-dose, post-dose (each cycle is 14 days), up to 24 months
Anti-drug Antibodies (ADA) for SKB264 and KL-A167 | Cycles 1-3, 5, 7, 9, and 11, every 6 cycles starting from Cycle 17 Day 1: within 1 h before infusion of SKB264 (each cycle is 14 days), up to 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu